CLINICAL TRIAL: NCT03405753
Title: Effects of Aronia Berry on Oxidative Stress, Cholesterol, Blood Pressure and Semen Quality
Brief Title: Potential Health Effects of Aronia Intake
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Odense University Hospital (Other)
Responsible Party: Principal Investigator, Jens Fedder, Professor, Odense University Hospital
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Prevention
Other Study IDs: Lab.Reprod.Biol.-Aronia
Record Dates: First submitted 2018-01-05; First posted 2018-01-23 (Actual); Last update posted 2023-11-03 (Actual); Status verified 2023-11

CONDITIONS: Health Effects of Aronia

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aroia (Active Comparator)
  Interventions: Dietary Supplement: Aronia, washout and then placebo; Dietary Supplement: Placebo, washout and then aronia
- Placebo (Placebo Comparator)
  Interventions: Dietary Supplement: Aronia, washout and then placebo; Dietary Supplement: Placebo, washout and then aronia

INTERVENTIONS:
Dietary Supplement: Aronia, washout and then placebo — Three tablets three times à day for three months then washout for three months, then three placebo tablets three times à day for three months. Blood samples and semen samples collected before and after each period of tablet intake.
Dietary Supplement: Placebo, washout and then aronia — Three tablets three times à day for three months, then washout for three months, then three aronia tablets three times à day for three months. Blood samples and semen samples collected before and after each period of tablet intake.

SUMMARY:
Intervention cross-over study during which participants receive standardized amounts of aronia berry tablets or placebo for three months, then wash out for three months, then aronia tablets or placebo for three months. The potential health effects are investigated. Following parameters are measured before and after each period of tablet intake: 1) Blood pressure, 2) Lipid fractions, 3) Testosterone, 4) Phase II markers, 5) HbA1c, 6) HSCRP, 7) F2-isoprostanes, and 8) semen quality.

ELIGIBILITY:
Inclusion Criteria:

* Healthy men with total cholesterol between 5 and 7 mmol/L, who do not take medication

Exclusion Criteria:

* Chronic diseases and intake of medication or antioxidants

Ages: 25 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 109 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2021-12-31 (Actual); Study Completion 2022-12-31 (Actual)

PRIMARY OUTCOMES:
Cholesterol | 9 months
  HDL, LDL and total cholesterol in mmol/L

SECONDARY OUTCOMES:
Phase II enzyme activity | 9 months
  Glutathion in U/mL
Phase II enzyme activity | 9 months
  Superoxid dismutase (SOD) in U/mL
Phase II enzyme activity | 9 months
  Catalase (CAT) in U/mL
Isoprostanes | 9 months
  Peroxidation of fatty acids measured in U/mL
Semen quality | 9 months
  Sperm count in million/mL
Semen quality | 9 months
  Motility in percent
Semen quality | 9 months
  DNA fragmentation in percent
Blood pressure | 9 months
  Systolic and diastolic blood pressure in mmHg
High Sensitivity C reactive protein | 9 months
  Acute phase reactant in mg/L

CONTACTS AND LOCATIONS:
Locations (1):
- Centre of Andrology & Fertility Clinic, Department D, Odense University Hospital, Odense, Denmark

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Sangild J, Faldborg A, Schousboe C, Fedder MDK, Christensen LP, Lausdahl AK, Arnspang EC, Gregersen S, Jakobsen HB, Knudsen UB, Fedder J. Effects of Chokeberries (Aronia spp.) on Cytoprotective and Cardiometabolic Markers and Semen Quality in 109 Mildly Hypercholesterolemic Danish Men: A Prospective, Double-Blinded, Randomized, Crossover Trial. J Clin Med. 2023 Jan 3;12(1):373. doi: 10.3390/jcm12010373. PMID 36615174